CLINICAL TRIAL: NCT00266084
Title: Double-Blinded Multicenter Clinical Study Assessing the Equivalence of the InPath Cervical Cell Collector to the Standard Endocervical Brush and Spatula in Patients Seeking Primary Pap Screening or Follow-up Screening
Brief Title: Clinical Trial for the Use of a Novel Cell Collector Device to Retrieve Cells From the Uterine Cervix
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Other Study IDs: 02-00-16
Record Dates: First submitted 2005-12-14; First posted 2005-12-15 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2001-11

CONDITIONS: Uterine Cervical Dysplasia; Uterine Cervical Intraepithelial Neoplasia; Uterine Cervical Neoplasia; Uterine Cervical Cancer
Keywords: Cervix; Uterus; Dysplasia; Cancer; Collector
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms; Neoplasms

SUMMARY:
This study tested the safety and performance of a new cell collector device and compared the results to those obtained with the current existing device that are being used routinely

DETAILED DESCRIPTION:
This study tested the feasibility, safety and efficacy of the new e2TM Collector, and compared its performance with the standard method for obtaining cervical cells for Pap test of endocervical cytobrush and Ayer's Spatula

ELIGIBILITY:
Inclusion Criteria:

Women ages >14 being followed for a previous abnormal Pap All patients will have signed an Informed Consent form prior to being enrolled in this study

Exclusion Criteria:

Patients who have had a hysterectomy

Min Age: 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85
Dates: Start 1999-08; Study Completion 2001-11

CONTACTS AND LOCATIONS:
Overall Officials: George I Gorodeski, MD PhD, Principal Investigator — University Hospitals of Cleveland, Case Western Reserve University